CLINICAL TRIAL: NCT00658112
Title: Measuring Adherence in Subjects With Acne Vulgaris in a Clinic Population Subtitle: Topical Benzoyl Peroxide for Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB0000027
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Benzoyl Peroxide 5% (Experimental): Subjects will be given standard instructions in the use of topical benzoyl peroxide gel and will be provided with a supply of medication fitted with a Medication Event Monitoring System (MEMS) cap. This cap records dates and times the assembly is opened which can be downloaded at the final visit and tabulated with associated software. When the tubes are weighed, data from the MEMS Caps will be collected. Study coordinators will record adherence, while assessors are blinded to adherence rates. All subjects will be assigned to treatment with topical benzoyl peroxide to the entire face.
  Interventions: Drug: Benzoyl Peroxide

INTERVENTIONS:
Drug: Benzoyl Peroxide — Benzoyl peroxide 5% gel. Applied once daily to face, minimum amount usable to cover area. Every day for six weeks.
  Other Names: Epiduo

SUMMARY:
The purpose of this research study is to see how often benzoyl peroxide is applied for acne. Use of medication was monitored electronically.

DETAILED DESCRIPTION:
We give subjects topical benzoyl peroxide, a standard first line acne treatment, in a container that records when the container is opened and closed. Subjects will simply be asked to "return in six weeks to see how well benzoyl peroxide works for them." Subjects initially will not be told that they are participating in a formal study. When they return with their medication, we will seek their informed consent to participate in the study. Verbal consent will be obtained at the beginning of the study. There will be no written consent obtained until the end of the study. By doing this, subjects will not be aware that adherence is being measured. Subjects will not be aware that they are participating in a study. Only if they consent would we then collect the medication container and monitor and retrieve the adherence data. If they do not consent, we will not have collected any research data on them except baseline acne severity measures which may have been collected anyway as part of their clinic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female 13 to 18 years of age with a diagnosis of mild to moderate acne vulgaris by a dermatologist will be eligible for participation.
* Verbal consent of participation must be given by parent or guardian and child.

Exclusion Criteria:

* Age less than 13 or greater than 18 years of age.
* Known allergy or sensitivity to topical benzoyl peroxide gel in the subject.
* Inability to complete all study-related visits.
* Introduction of any other prescription medication, topical or systemic, for acne vulgaris while participating in the study.
* Subjects should not be using topical retinoids or benzoyl peroxide products, including Proactive® or topical prescription medications for the treatment of acne vulgaris for at least 2 weeks prior to beginning the study. Oral medications for the treatment of acne should not have been used at least 4 weeks prior to beginning the study.
* Women that are actively trying to become pregnant or wish to become pregnant during the time frame the study is to take place will be excluded.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Benzoyl Peroxide 5%
Started | 20
Completed | 11
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Benzoyl Peroxide 5%
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Adherence to medication use as measured by MEMS cap reported as % of prescribed doses actually applied
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: percentage of doses actually applied
Arm/Group | Benzoyl Peroxide 5%
Number analyzed (Participants) | 11
percentage of doses actually applied | 46.5 [14 to 79]

ADVERSE EVENTS:
Arm/Group | Benzoyl Peroxide 5%
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes